CLINICAL TRIAL: NCT04264039
Title: Anti-CD19 Universal CAR-T Cells for CD19+ B Cell Hematologic Malignancies: a Multi-center, Uncontrolled Trial
Brief Title: Anti-CD19 U-CAR-T Cell Therapy for B Cell Hematologic Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry); 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Central South University (Other); First Affiliated Hospital of Kunming Medical University (Other); The General Hospital of Western Theater Command (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Nanfang Hospital, Southern Medical University (Other); Fujian Medical University Union Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Xi Zhang, MD, Chef of Hematology Department, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: antiCD19-UCAR-T
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; B-cell Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, B-Cell | interventions — fludarabine; Cyclophosphamide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19 UCAR-T cells (Experimental): After preconditioning with chemotherapy ( Fludarabine, Cytoxan and/or Melphalan), the dosage of anti-CD19 UCAR-T cells between 1 and 5 ×10^7 cells/Kg will be evaluated
  Interventions: Biological: anti-CD19 UCAR-T cells; Drug: Fludarabine; Drug: Cytoxan; Drug: Melphalan

INTERVENTIONS:
Biological: anti-CD19 UCAR-T cells — Dose range:1 to 5 ×10^7 cells/Kg, Dose level one: 1×10^7 cells/Kg, Dose level two: 3×10^7 cells/Kg, Dose level three:5 ×10^7 cells/Kg
Drug: Fludarabine — 30mg/m^2 per day for 6 days
Drug: Cytoxan — 300mg/m^2 per day for 2 to 6 days determined by tumor burden at baseline
Drug: Melphalan — 50 to 70 mg/m^2 in total for 1 or 2 days, whether to use determined by tumor burden at baseline

SUMMARY:
The stunning response rate of anti-CD19(cluster of differentiation antigen 19) auto-CAR(chimeric antigen receptor)-T cell therapy brings hope to patients with relapsed or refractory B-cell hematologic malignancies. However, based on open clinical trials, using patients' T cells might encounter the failure of apheresis available T cells, even if successful, the time needed for the manufacture could also cause the irreversible disease progress. Furthermore, the cost of auto-CAR-T cells is not affordable for most patients. So to provide an accessible and affordable anti-CD19 CAR-T cell therapy for patients with B-cell hematologic malignancies, we launch such a trial that using the edited T cells from healthy donors to manufacture universal CAR-T cells and adapt it in patients with CD19+ B-cell leukemia or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of recurrent B-cell acute lymphoblastic leukemia (B-ALL), B-cell acute lymphoblastic lymphoma (B-LLy), or B-non-Hodgkin lymphoma (B-NHL)

  2. CD19-positive tumor (≥20% CD19 positive blasts by flow cytometry or immunohistochemistry (tissue)）

  3. Hgb ≥ 7.0 (can be transfused)

  4. Life expectancy greater than 12 weeks

  5. Informed consent explained to, understood by and signed by the patient/guardian. The patient/guardian is given a copy of informed consent.

Exclusion Criteria:

1. Pregnant or lactating.
2. Tumor in a location where enlargement could cause airway obstruction (per investigator discretion).
3. Active infection with HIV or HTLV.
4. Clinically significant viral infection or uncontrolled viral reactivation of EBV(Epstein-Barr virus), CMV(cytomegalovirus), ADV(adenovirus), BK-virus, or HHV(human herpesvirus)-6.
5. Any of the following cardiac criteria: Atrial fibrillation/flutter; Myocardial infarction within the last 12 months; Prolonged QT syndrome or secondary prolonged QT, per investigator discretion. Cardiac echocardiography with LVSF (left ventricular shortening fraction)<30% or LVEF(left ventricular ejection fraction)<50%; or clinically significant pericardial effusion. Cardiac dysfunction NYHA(New York Heart Association) III or IV (Confirmation of absence of these conditions on echocardiogram within 12 months of treatment).
6. CNS abnormalities: Presence of CNS(central nervous system)-3 disease defined as detectable cerebrospinal blast cells in a sample of CSF(cerebrospinal fluid) with ≥ 5 WBC( white blood cell)s per mm3 (unless negative by the Steinherz/Bleyer algorithm); Presence of any CNS disorder such as an uncontrolled seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
the anti-tumor efficiency of anti-CD19 UCAR-T cells | 4 weeks after infusion
  ratio of bone marrow blast cells and/or the measurable lesion size and strandralized uptake value

SECONDARY OUTCOMES:
the long-term efficiency of anti-CD19 UCAR-T cells | 3 and 6 months after infusion
  ratio of bone marrow blast cells and/or the measurable lesion size and strandralized uptake value

CONTACTS AND LOCATIONS:
Overall Officials: Xi Zhang, MD, Principal Investigator — Xinqiao Hospital of Chongqing
Locations (1):
- Department of Hematology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China